CLINICAL TRIAL: NCT00243750
Title: Open Study for the Evaluation of the Efficacy of Methotrexate 20mg Given Subcutaneously in Patients With Active Ankylosing Spondylitis
Brief Title: Methotrexate in Ankylosing Spondylitis (MTX in AS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: MTX-01
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2005-12-09 (Estimated); Status verified 2003-08

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; trial; methotrexate
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Methotrexate

INTERVENTIONS:
Drug: Methotrexate

SUMMARY:
Assessing the efficacy and tolerability of methotrexate 15mg sc in the first month of treatment- if well tolerated methotrexate 20mg sc in the following 3 months in patients with active anklyosing spondylitis

DETAILED DESCRIPTION:
Ankylosing spondylitis is an inflammatory rheumatic disease mit main affection of the spine. However peripheral joints, entheses and the eyes can also be affected. The rheumatic symptoms of the patients typically show good response to nonsteroidal antirheumatic drugs.

In contrast to rheumatoid arthritis in ankylosing spondylitis there is no evidence that therapy with disease modifying antirheumatic drugs is effective (DMARD). Next to studies with the DMARD sulfasalazine, which seems to be effective mainly in peripheral joint involvement and in which a possible effect in short disease duration also seems to exist for axial involvement, in regards of other DMARDs there are only small studies or case reports.

In terms of methotrexate only small studies with a dosage of 7,5mg - 10 mg - maximally 15mg (perorally in single patients) have been published. In three open studies in 11- 34 patients treated with methotrexate 7,5mg - maximally 15mg perorally over a time duration of 24 weeks until maximally 3 years there a certain effectiveness partly in spinal symptoms, partly in peripheral joint involvement (1, 2, 3). In both double blind controlled studies with 30 and 50 patients respectively with a dosage of 7,5 and 10mg methotrexate respectively no significant effectiveness was shown (4,5). To summarize, in the different studies no effectiveness could be shown clearly.

Therapy with methotrexate in patients with inflammatory rheumatic diseases - especially in rheumatoid arthritis- belongs to standard therapy. In Germany methotrexate is given in about 70% of cases because of its good effectiveness as therapy of first choice. In the treatment of psoriatic arthritis representing a disease which is similar to ankylosing spondylitis in regards to pathogenesis, methotrexate therapy could be established in a dosage of 20mg parenterally and 25mg perorally respectively successfully. Bearing this in mind it is even more surprising that there are no data about methotrexate in this dosages for the treatment of ankylosing spondylitis. According to the German rheumatic register (so-called "rheumatologische Kerndokumentation", PD. Dr. A. Zink, DRFZ, Berlin) already about 20% of patients with ankylosing spondylitis are treated with methotrexate by German rheumatologists. For this reason it is makes sense to perform a study for the treatment of patients with active ankylosing spondylitis with methotrexate in a dosage of 20mg. In the therapy of rheumatoid arthritis a combination of methotrexate and TNFalpha blocking agents leads to an enhancement of effectiveness and reduction of side effects. For this reason the effectivenss of methotrexate in ankylosing spondylitis is also very interesting in regards to a possible combination with TNFalpha blocking agents which have shown to be very successful in the treatment of ankylosing spondyltitis.

ELIGIBILITY:
Inclusion criteria:

* Definite ankylosing spondylitis according to the New York criteria of 1984.
* Known ankylosing spondylitis according to the modified New York criteria from 1984
* age 18- 70 years
* insufficient therapy with nonsteroidal antirheumatic drugs
* BASDAI > 4
* therapy with DMARD (sulfasalazine, hydroxychloroquine, leflunomide, methotrexate ≤ 10 mg etc.) allowed before study start if discontinued at least 1 month before study start; elimination of leflunomide with colestyramin of coal if necessary. · therapy with biologics (TNF-alpha blocking agents, IL-1-blocking agents etc.) discontinued at least 3 months before study start
* therapy with steroids ≤ 10 mg at least 4 weeks stable before study start
* patient should be willing to prevent pregnancy by using accepted contraceptive methods until the end of study
* signed informed consent
* patient should be able to administer study drug
* exclusion of pregnancy in female patients with childbearing potential

Exclusion criteria:

* intake of glucocorticosteroids of > 10 mg, therapy with intraarticular steroids within last 4 weeks before study start
* previous therapy with methotrexate > 10 mg
* allergy to methotrexate or parts of medication
* pregnancy/ lactation
* current severe infections, suspicion for opportunistic infections (Herpes zoster, cytomegaly-, pneumocystis carinii-infection) or within the last 4 months , HIV- infection
* malignant disease within the last 5 years
* severe cardiac, renal, hematologic, endocrine, pulmonary, neurological, gastrointestinal (e.g. gastroesophageal ulcer) or hepatic (viral hepatitis, toxic liver disease etc.) disease, uncontrolled high blood pressure, recurrent thrombosis/ emboly, significant disease in hematopoesis.
* active immunization within last 4 weeks or immunization which is planned for study time
* significant findings in the laboratory: hemoglobin < 8,5 mg/dl, leukopenia < 3,5 /nl, thrombopenia< 100 /nl, creatinine>200 µmol/l, liver enzymes or alkaline phosphate > 1,5-fold over upper limit of normal
* significant pathologic findings in physical examination
* particpation in another clinical trial in last 30 days
* substance abuse, e.g. cocaine, heroine, alcohol abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-09; Study Completion 2005-11

PRIMARY OUTCOMES:
improvement of disease activity parameters according to ASAS - 20% response

SECONDARY OUTCOMES:
improvement of BASDAI, of pain on a scale from 0-10, reduction of CRP/ ESR (inflammatory serum parameters), reduction of BASFI, BASMI, number of swollen and tender joints, number of enthesitic locations, improvement of life quality.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Sieper, Prof., Principal Investigator — Charité Campus Benjamin-Franklin, Rheumatology
Locations (1):
- Charité Campus Benjamin-Franklin, Rheumatology, Berlin, Germany